CLINICAL TRIAL: NCT03302533
Title: Can Secondary Total Elbow Arthroplasty After Failed Internal Fixation or Non-operative Treatment of Distal Humeral Fractures Achieve Equal Results as Primary Arthroplasty?
Status: Completed | Type: Observational
Sponsor: Diakoniekrankenhaus Friederikenstift (Other)
Responsible Party: Principal Investigator, Dr. Alexander Ellwein, Assistant Physician, Diakoniekrankenhaus Friederikenstift
Other Study IDs: 001-2017
Record Dates: First submitted 2017-09-30; First posted 2017-10-05 (Actual); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Elbow Fracture; Elbow Arthropathy
Keywords: distal humerus fracture; total elbow arthroplasty; elbow prosthesis; delayed arthroplasty; revision surgery
MeSH Terms: conditions — Elbow Fractures; Humeral Fractures, Distal | interventions — Arthroplasty, Replacement, Elbow

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary arthroplasty: All patients who received TEA for an acute trauma with fracture of the distal humerus.
  Interventions: Procedure: Total elbow arthroplasty
- Secondary arthroplasty: All patients who received TEA due to a failed reconstruction or non-operative treatment after a distal humerus fracture.
  Interventions: Procedure: Total elbow arthroplasty

INTERVENTIONS:
Procedure: Total elbow arthroplasty — Implantation of a total elbow arthroplasty after distal humerus fracture

SUMMARY:
Total elbow arthroplasty (TEA) results in immediate pain release with good functional results after distal humerus fractures. But still open reduction and internal fixation is recommended as treatment of choise due to a lifelong loading limitiation, unknown implant survival and problematic revision surgery after TEA. The purpose of this study was to compare functional results and complication rates after primary total elbow arthroplasty (TEA) and TEA after failed reconstruction or non-operative treatment (secondary TEA) in the treatment of distal humerus fractures. We hypothesised that clinical and functional results are better for primary TEA with less complications.

DETAILED DESCRIPTION:
Total elbow arthroplasty (TEA) results in immediate pain release with good functional results after distal humerus fractures. But still open reduction and internal fixation is recommended as treatment of choise due to a lifelong loading limitiation, unknown implant survival and problematic revision surgery after TEA. The purpose of this study was to compare functional results and complication rates after primary total elbow arthroplasty (TEA) and TEA after failed reconstruction or non-operative treatment (secondary TEA) in the treatment of distal humerus fractures.

This retrospective study was performed at a level I trauma centre. All patients were informed about the study and provided written informed consent.

All patients undergoing total elbow arthroplasty (TEA) were identified by electronically screening our database by the OPS codes 5-824.4 (implantation of a linked TEA) and 5-824.5 (implantation of an unlinked TEA) between August 2008 and May 2014. Based on patient records and x-rays the indication for implantation of the TEA was retrospectively reviewed. All patients, who received a TEA for an acute trauma with fracture of the distal humerus (primary TEA) or due to a failed reconstruction or non-operative treatment after a distal humerus fracture (secondary TEA), were included in this study. A minimum follow-up of 6 months was set as inclusion criterion. Exclusion criteria were previous injury at the fractured elbow, neuro-muscular disease, cortisone or other immune suppressive therapy and open fracture grade II or higher according to Tscherne and Ostern.The patient records were reviewed for demographic and perioperative data. If the initial treatment was not conducted in our department, radiographs and patient records were requested. The follow-up examination included the evaluation of the range of motion and stability of the elbow, actual pain and satisfaction of the patient. To objectify the functional result the Mayo Elbow Performance Score (MEPS) and Disabilities of the Arm, Shoulder and Hand Score (DASH) were determined. Additionally, complications and revision surgeries were recorded. Complications were split up into minor (nerve irritation or postoperative haematoma) and major complications, which required a revision of the prosthesis. Periprosthetic fractures due to renewed fall with an adequate trauma were not counted as complication.

Perioperative data, the functional result (range of motion, MEPS, DASH) and postoperative complications were described for each group. Subsequently, these results were statistically compared using the Mann-Whitney U test as a two-way analysis of variance for independent factors. A p-value ≤ 0.05 was considered statistically significant. The statistical analysis was performed using SPSS for MAC (IBM SPSS Statistics 22, Chicago, Illinois).

We hypothesised that clinical and functional results are better for primary TEA with less complications.

ELIGIBILITY:
Minimum age: 18 years Sex: All

Inclusion Criteria:

* Total elbow arthroplasty for an acute trauma with fracture due to an acute trauma
* Total elbow arthroplasty due to failed reconstruction after distal humerus fracture
* Total elbow arthroplasty after non-operatic treatment after distal humerus fracture

Exclusion Criteria:

* previous injury at the fractured elbow
* neuro-muscular disease
* cortisone or other immune suppressive therapy
* open fracture grade II or higher according to Tscherne and Ostern

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Out of 35 patients, who fit the inclusion criteria, six had died from unrelated causes. 23 patients participated in the study, since six patients were lost to follow-up. Nine of the 23 patients (mean age: 70 years; 8 women) had implantation of a primary TEA. The remaining 14 patients (mean age: 63 years; 11 women) received secondary implantation of a TEA. The secondary TEA was implanted after an implant failure in four patients, twice because of a non-union (one after reconstruction and one after non-operative therapy), and in three patients because of a non-union with an additional partial necrosis of the distal humerus. Two patients received secondary TEA because of a posttraumatic arthritis after internal fixation and three times because of a posttraumatic arthritis after non-operative treatment. The mean follow-up was 28 months (range: 6 - 73) with a mean age of 66 years (range: 41 - 85).
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2013-01-21 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Range of motion | minimum follow-up: 6 months
  Measurement of the range of motion for extension/flexion
Mayo Elbow Performance Score | minimum follow-up: 6 months
  Objective score evaluation the function of the elbow

SECONDARY OUTCOMES:
Complication | minimum follow-up: 6 months
  appearance of a complication

OTHER OUTCOMES:
DASH score | minimum follow-up: 6 months
  Disabilities of the Arm, Shoulder and Hand: subjective score evaluation the function

IPD SHARING:
Plan to Share IPD: No